CLINICAL TRIAL: NCT04865991
Title: Comparison of Propofol Target Controlled Infusion (TCI) and Sevoflurane Recovery Time in Vitrectomy Surgery: a Randomized Controlled Trial
Brief Title: Comparison of Propofol Target Controlled Infusion (TCI) and Sevoflurane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Aida Rosita Tantri, MD, Indonesia University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IndonesiaUAnes101
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Vitreous Detachment
Keywords: vitrectomy; propofol; sevoflurane; TCI
MeSH Terms: conditions — Vitreous Detachment | interventions — Sevoflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TCI propofol group (Experimental): Subjects in the TCI propofol group received TCI propofol for anesthesia maintenance, Ce value was titrated until a targeted BIS score of 40-60 achieved.
  Interventions: Procedure: TCI Propofol
- sevoflurane group (Active Comparator): Subjects in the sevoflurane group received sevoflurane 2 volume%, which were titrated up/down every 5 minutes to get a targeted BIS score of 40-60.
  Interventions: Procedure: Sevoflurane

INTERVENTIONS:
Procedure: TCI Propofol — Peripheral venous catheters were placed in all subjects. Subjects in the TCI propofol group had one specific intravenous catheter for propofol infusion apart from medication or intravenous fluid line. Subjects in the TCI Propofol group received TCI propofol (Schneider) with targeted Ce 4 -5 mcg/ml for anesthesia induction and maintenance. Subjects in the TCI propofol group received TCI propofol for anesthesia maintenance, Ce value was titrated until a targeted BIS score of 40-60 achieved.
  Arms: TCI propofol group
Procedure: Sevoflurane — subjects in the sevoflurane group were cannulated only with one venous catheter. Midazolam 0.05 mg/kg BW and fentanyl 1 mcg/kg BW were given as premedication. Subjects in the sevoflurane group received intravenous propofol 1 - 2 mg/kg BW.
  Arms: sevoflurane group

SUMMARY:
This study was an experimental, single-blinded, randomized controlled trial that aimed to compare recovery time between TCI propofol and sevoflurane. After ethical approval from Research Ethical Committee Faculty of Medicine, Universitas Indonesia (879/UN2.F1/ETIK/2017) and informed consent, patients aged 18-65 years old, body mass index 18 - 30 kg/m2, American Society of Anesthesiologists (ASA) status I-II who were scheduled for vitrectomy surgery under general anesthesia, at Kirana's Eye Operating Theatre Cipto Mangunkusumo National Referral Hospital from September until December 2017, were recruited in this study. All subjects would be recruited with a consecutive sampling method and randomly assigned into two groups, the TCI propofol group and sevoflurane group. Block random allocation was done for all subjects by using the random allocator program Winpepi.

DETAILED DESCRIPTION:
This study was an experimental, single-blinded, randomized controlled trial that aimed to compare recovery time between TCI propofol and sevoflurane. After ethical approval from Research Ethical Committee Faculty of Medicine, Universitas Indonesia (879/UN2.F1/ETIK/2017) and informed consent, patients aged 18-65 years old, body mass index 18 - 30 kg/m2, American Society of Anesthesiologists (ASA) status I-II who were scheduled for vitrectomy surgery under general anesthesia, at Kirana's Eye Operating Theatre Cipto Mangunkusumo National Referral Hospital from September until December 2017, were recruited in this study. Patients with hemodynamic instability, allergy, raised intracranial pressure, and a history of hyperthermia malignant, were excluded from this study. Patients who have hearing disturbance, history of alcohol, opioid, or psychotropic drugs consumption before surgery, suffered from neuropsychiatric disease, and electrolyte imbalance was also excluded from this study. Patients who experience intraoperative cardiorespiratory disturbance, surgery duration less than 35 minutes or more than 3 hours and 30 minutes, and patients with temperature abnormalities before being extubated from LMA would be excluded from the trial.

Sample size The sample size calculation was performed with the unpaired numerical analytic equation. At least eighteen subjects for each group should include in this study. With the ten percent dropout possibility, twenty subjects will be recruited for each group, resulting in a total sample size of 40 subjects. All subjects would be recruited with a consecutive sampling method and randomly assigned into two groups, the TCI propofol group and sevoflurane group. Block random allocation was done for all subjects by using the random allocator program Winpepi.

Study Protocols Peripheral venous catheters were placed in all subjects. Subjects in the TCI propofol group had one specific intravenous catheter for propofol infusion apart from medication or intravenous fluid line. In comparison, subjects in the sevoflurane group were cannulated only with one venous catheter. Midazolam 0.05 mg/kg BW and fentanyl 1 mcg/kg BW were given as premedication. Subjects in the TCI Propofol group received TCI propofol (Schneider) with targeted Ce 4 -5 mcg/ml for anesthesia induction and maintenance. Subjects in the sevoflurane group received intravenous propofol 1 - 2 mg/kg BW. BIS scores in both groups was titrated down to 50. Laryngeal mask no.3 or no.4 was inserted three minutes after administering atracurium 0.25 mg/kg BW. All subjects were ventilated with tidal volume 8 ml/kg BW, 12 times/minutes, oxygen fraction 50%.

Subjects in the TCI propofol group received TCI propofol for anesthesia maintenance, Ce value was titrated until a targeted BIS score of 40-60 achieved. Subjects in the sevoflurane group received sevoflurane 2 volume%, which were titrated up/down every 5 minutes to get a targeted BIS score of 40-60. Blood pressure, heart rate, oxygen saturation, and BIS score were monitored every 5 minutes. Fentanyl 1 mcg/ kg BW was added if there was an increase in blood pressure, heart rate and or BIS score that couldn't be overcome by increasing the dose of TCI propofol or sevoflurane.

Surgery was considered done when the palpebral retractor had been removed. After spontaneous ventilation reverted, neostigmine 0.04 mg/kg BW and atropine 0.04 mg/kg BW as a reversal agent were given. Laryngeal mask was removed when the anesthesia still deep enough and subjects were monitored afterward. Time when TCI propofol and sevoflurane were discontinued was recorded (T0). Time when the patient was fully awake and could follow simple orders such as raising hands was recorded (Tp). Recovery time was the duration from T0 to Tp. Unwanted events during recovery, such as agitation and nausea-vomiting were recorded. Total fentanyl usage during surgery was also recorded. Statistical analysis was performed using Statistical Product for Social Sciences (SPSS) software 21.0 for windows. T-Test or Mann-Whitney analysis was done depending on the data normality test.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-65 years old
* body mass index 18 - 30 kg/m2
* American Society of Anesthesiologists (ASA) status I-II
* scheduled for vitrectomy surgery under general anesthesia

Exclusion Criteria:

* Patients with hemodynamic instability, allergy, raised intracranial pressure, and a history of hyperthermia malignant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Recovery time | 2 hour
  Recovery time was the duration from T0 to Tp. Unwanted events during recovery, such as agitation and nausea-vomiting were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Cental National Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No